CLINICAL TRIAL: NCT00624468
Title: A Two-arm, Randomized, Double-blind, Placebo-controlled, Multicenter Phase II Study to Evaluate Safety and Tolerability and to Explore the Neuroprotective Effect of Atacicept as Assessed by Optical Coherence Tomography (OCT) in Subjects With Optic Neuritis (ON) as Clinically Isolated Syndrome (CIS) Over a 36-week Treatment Course
Brief Title: Atacicept in Subjects With Optic Neuritis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: EMD Serono voluntarily decided to terminate this trial after observing increased MS disease activity in trial 28063 ATAMS [Please refer to ATAMS]
Sponsor: EMD Serono (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 28156
Record Dates: First submitted 2008-02-15; First posted 2008-02-27 (Estimated); Results first posted 2016-02-17 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-01

CONDITIONS: Optic Neuritis
Keywords: atacicept; neuritis
MeSH Terms: conditions — Optic Neuritis; Neuritis | interventions — TACI receptor-IgG Fc fragment fusion protein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atacicept (Experimental)
  Interventions: Drug: Atacicept
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo matched to atacicept

INTERVENTIONS:
Drug: Atacicept — Atacicept will be administered subcutaneously at a dose of 150 milligram (mg) twice a week for initial 4 weeks as loading dose, followed by 150 mg once a week for subsequent 32 weeks.
  Arms: Atacicept
Drug: Placebo matched to atacicept — Placebo matched to atacicept will be administered subcutaneously twice a week for initial 4 weeks, followed by once a week for subsequent 32 weeks.
  Arms: Placebo

SUMMARY:
This study was intended to evaluate the efficacy, safety and tolerability of atacicept compared to placebo and to explore the neuroprotective effect of atacicept as assessed by OCT in subjects with ON as CIS. The study was randomized. Study medication was administered via subcutaneous (under the skin) injections.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of unilateral symptomatic optic neuritis as first clinical manifestation within 28 days between onset of symptoms and study Day 1
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Pre treatment with immunosuppressants and immunomodulating drugs
* Relevant cardiac, hepatic and renal diseases
* Clinical significant abnormalities in blood cell counts and immunoglobulin levels
* Clinical significant acute or chronic infections
* Other protocol defined exclusion criteria could apply

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2008-06; Primary Completion 2009-09 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — EMD Serono, an affiliate of MerckKGaA, Darmstadt, Germany
Locations (28):
- United States (8):
  - Research Site, Birmingham, Alabama
  - Research Site, Aurora, Colorado
  - Research Site, Fairfield, Connecticut
  - Research Site, Jacksonville, Florida
  - Research Site, East Lansing, Michigan
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Houston, Texas
  - Research Site, Burlington, Vermont
- Research Site, Parkville, Victoria, Australia
- Research Site, Brussels, Belgium
- Canada (3):
  - Research Site, Vancouver, British Columbia
  - Research Site, Ottawa, Ontario
  - Research Site, Montreal, Quebec
- Czechia (2):
  - Research Site, Hradec Králové
  - Research Site, Olomouc
- Research Site, Paris, France
- Germany (4):
  - Research Site, Freiburg im Breisgau
  - Research Site, Munich
  - Research Site, Tübingen
  - Research Site, Würzburg
- Lebanon (2):
  - Research Site, Beirut
  - Research Site, Dbaïyé
- Spain (3):
  - Research Site, Barcelona
  - Research Site, Seville
  - Research Site, Valencia
- Research Site, Lausanne, Switzerland
- United Kingdom (2):
  - Research Site, London
  - Research Site, Sheffield

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Double-blind Period: Placebo matched to atacicept was administered subcutaneously twice a week for initial 4 weeks, followed by once a week for subsequent 32 weeks.
- Atacicept: Double-blind Period: Atacicept was administered subcutaneously at a dose of 150 milligram (mg) twice a week for initial 4 weeks as loading dose, followed by 150 mg once a week for subsequent 32 weeks.
- Placebo: SFU Period: Subjects who received placebo matched to atacicept in double-blind period were included in safety follow-up (SFU) period (60 weeks) following premature termination of the trial.
- Atacicept: SFU Period: Subjects who received atacicept in double-blind period were included in SFU period (60 weeks) following premature termination of the trial.
Period: Double-blind Period
Arm/Group | Placebo: Double-blind Period | Atacicept: Double-blind Period | Placebo: SFU Period | Atacicept: SFU Period
Started | 17 | 17 | 0 | 0
Completed | 3 | 4 | 0 | 0
Not Completed | 14 | 13 | 0 | 0
Not completed — Early Termination Initiated by Sponsor | 13 | 12 | 0 | 0
Not completed — Withdrew Prematurely | 1 | 1 | 0 | 0
Period: Safety Follow-up (SFU) Period
Arm/Group | Placebo: Double-blind Period | Atacicept: Double-blind Period | Placebo: SFU Period | Atacicept: SFU Period
Started | 0 | 0 | 13 | 14
Completed | 0 | 0 | 11 | 11
Not Completed | 0 | 0 | 2 | 3
Not completed — Lost to Follow-up | 0 | 0 | 1 | 2
Not completed — Other | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo: Double-blind Period | Atacicept: Double-blind Period | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.3 (7.1) | 30.6 (10.2) | 31.4 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 27
  Male | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Retinal Nerve Fiber Layer (RNFL) Thickness in the Affected Eye at Last Observed Value (LOV)
Description: The RNFL thickness was measured for 12 sectors (every 30 degrees) per eye in triplicate by optical coherence tomography (OCT) measurements and were then averaged over 12 sectors. The change in RNFL thickness at LOV visit was calculated as RNFL thickness at LOV minus RNFL thickness at baseline.
Time Frame: Baseline, LOV (Week 48)
Population: ITT population included all randomized participants. Here, "n" signifies those participants who were evaluable for the specified category.
Measure: Mean (Standard Deviation); unit: micrometer
Groups:
- Atacicept: Double-blind Period: Atacicept was administered subcutaneously at a dose of 150 mg twice a week for initial 4 weeks as loading dose, followed by 150 mg once a week for subsequent 32 weeks.
Arm/Group | Placebo: Double-blind Period | Atacicept: Double-blind Period
Number analyzed (Participants) | 17 | 17
micrometer
  Baseline (n = 17, 17) | 103.893 (17.271) | 104.170 (8.832)
  Change at LOV (n = 16, 15) | -17.317 (15.158) | -8.636 (10.056)

2. Secondary Outcome: Difference in Retinal Nerve Fibre Layer (RNFL) Thickness Between the Affected Eye and Fellow Eye
Description: The RNFL thickness was measured for 12 sectors (every 30 degrees) per eye in triplicate by optical coherence tomography (OCT) measurements and was then averaged over 12 sectors. Difference was calculated as RNFL thickness in affected eye minus RNFL thickness in fellow eye.
Time Frame: Weeks 12, 24 and 36
Population: ITT population included all randomized participants. Here, "N" (number of participants analyzed) signifies those participants who were evaluable for this outcome measure and "n" signifies those participants who were evaluable for the specified category.
Measure: Mean (Standard Error); unit: micrometer
Arm/Group | Placebo: Double-blind Period | Atacicept: Double-blind Period
Number analyzed (Participants) | 13 | 13
micrometer
  Change at Week 12 (n = 13, 13) | -14 (4) | -7.9 (1.5)
  Change at Week 24 (n = 4, 5) | -7 (6.9) | -10.6 (3.7)
  Change at Week 36 (n = 3, 4) | -7.5 (8.8) | -9.4 (6.6)

3. Secondary Outcome: Change From Baseline in Retinal Nerve Fiber Layer (RNFL) Thickness in the Affected Eye at Weeks 12 and 24
Description: The RNFL thickness was measured for 12 sectors (every 30 degrees) per eye in triplicate by OCT measurements and was then averaged over 12 sectors. The change in RNFL thickness at Weeks 12 and 24 was calculated as RNFL thickness at Weeks 12 and 24 minus RNFL thickness at baseline, respectively.
Time Frame: Baseline, Weeks 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: micrometer
Arm/Group | Placebo: Double-blind Period | Atacicept: Double-blind Period
Number analyzed (Participants) | 13 | 13
micrometer
  Baseline (n=17, 17) | 103.893 (17.271) | 104.170 (8.832)
  Change at Week 12 (n = 13, 13) | -17.036 (13.919) | -9.356 (9.532)
  Change at Week 24 (n = 4, 5) | -17.815 (16.505) | -11.234 (14.230)

4. Secondary Outcome: Change From Baseline in Macular Thickness at 3 Millimeter (mm) Around Fovea in the Affected Eye at Weeks 12, 24 and 36
Description: The change in macular thickness at 3 mm around fovea in the affected eye at Weeks 12, 24 and 36 was calculated as macular thickness at 3 mm in the affected eye at Weeks 12, 24 and 36 minus macular thickness at 3 mm in the affected eye at baseline, respectively.
Time Frame: Baseline, Weeks 12, 24 and 36
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: micrometer
Arm/Group | Placebo: Double-blind Period | Atacicept: Double-blind Period
Number analyzed (Participants) | 17 | 17
micrometer
  Baseline (n = 17, 17) | 1054.4 (76.5) | 1070.6 (72.7)
  Change at Week 12 (n = 13, 13) | -29.3 (34.4) | -34.0 (21.8)
  Change at Week 24 (n = 4, 5) | -72.5 (47.0) | -50.4 (47.7)
  Change at Week 36 (n = 3, 4) | -32.7 (30.7) | -40.0 (51.3)

5. Secondary Outcome: Change From Baseline in Macular Thickness at 6 Millimeter (mm) Around Fovea in the Affected Eye at Weeks 12, 24 and 36
Description: The change in macular thickness at 6 mm around fovea in the affected eye at Weeks 12, 24 and 36 was calculated as macular thickness at 6 mm in the affected eye at Weeks 12, 24 and 36 minus macular thickness at 6 mm in the affected eye at baseline, respectively.
Time Frame: Baseline, Weeks 12, 24 and 36
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: micrometer
Arm/Group | Placebo: Double-blind Period | Atacicept: Double-blind Period
Number analyzed (Participants) | 17 | 17
micrometer
  Baseline (n = 17, 17) | 954.4 (57.4) | 947.5 (61.3)
  Change at Week 12 (n = 13, 13) | -36.1 (28.4) | -32.8 (25.2)
  Change at Week 24 (n = 4, 5) | -63.8 (32.7) | -46.2 (36.5)
  Change at Week 36 (n = 3, 4) | -33.3 (33.7) | -34.8 (46.0)

6. Secondary Outcome: Change From Baseline in Macular Volume in the Affected Eye at Weeks 12, 24 and 36
Description: The change in macular volume in the affected eye at Weeks 12, 24 and 36 was calculated as macular volume in the affected eye at Weeks 12, 24 and 36 minus macular volume in the affected eye at baseline, respectively.
Time Frame: Baseline, Weeks 12, 24 and 36
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cubic micrometer
Arm/Group | Placebo: Double-blind Period | Atacicept: Double-blind Period
Number analyzed (Participants) | 17 | 17
cubic micrometer
  Baseline (n = 17, 17) | 6.8865 (0.4199) | 6.8794 (0.4372)
  Change at Week 12 (n = 13, 13) | -0.2389 (0.1991) | -0.2301 (0.1612)
  Change at Week 24 (n = 4, 5) | -0.4630 (0.2466) | -0.3292 (0.2674)
  Change at Week 36 (n = 3, 4) | -0.2353 (0.2253) | -0.2533 (0.3205)

7. Secondary Outcome: Low-Contrast Letter Acuity: Total Number of Letters Correctly Identified
Description: Low-contrast letter acuity was measured by using the Sloan Charts at 1.25 fraction (%) and 2.5%. Sloan letters are a set of optotypes used to test visual acuity. Total number of letters correctly identified in the affected and fellow eye were reported. The possible Sloan Chart range is 0 to 70. More the number of letters identified, better is the visual acuity.
Time Frame: Weeks 12, 24 and 36
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Placebo: Double-blind Period | Atacicept: Double-blind Period
Number analyzed (Participants) | 15 | 14
letters
  Sloan chart 1.25%, affected eye: Week 12 (n=15,14) | 14.7 (14.7) | 15.7 (19.0)
  Sloan chart 1.25%, affected eye: Week 24 (n = 5,5) | 16.2 (13.6) | 13.4 (18.4)
  Sloan chart 1.25%, affected eye: Week 36 (n = 3,4) | 24.7 (8.1) | 9.8 (18.8)
  Sloan chart 2.5%, affected eye: Week 12 (n=15, 14) | 25.6 (16.7) | 22.1 (19.5)
  Sloan chart 2.5%, affected eye: Week 24 (n = 5, 5) | 26.8 (15.2) | 21.4 (19.3)
  Sloan chart 2.5%, affected eye: Week 36 (n = 3, 4) | 38.7 (4.7) | 20.3 (18.7)
  Sloan chart 1.25%, fellow eye: Week 12 (n=15,14) | 25.7 (13.1) | 25.9 (16.5)
  Sloan chart 1.25%, fellow eye: Week 24 (n = 5,5) | 22.2 (16.1) | 24.6 (18.4)
  Sloan chart 1.25%, fellow eye: Week 36 (n = 3,4) | 35.3 (4.2) | 19.8 (20.6)
  Sloan chart 2.5%, fellow eye: Week 12 (n=15, 14) | 35.3 (13.4) | 36.4 (12.7)
  Sloan chart 2.5%, fellow eye: Week 24 (n = 5, 5) | 33.6 (18.2) | 35.8 (15.4)
  Sloan chart 2.5%, fellow eye: Week 36 (n = 3, 4) | 45.7 (4.5) | 32.5 (19.1)

8. Secondary Outcome: Contrast Sensitivity: Total Number of Letters Correctly Identified
Description: Contrast Sensitivity was measured using the Pelli-Robson Charts. Pelli-Robson chart is used for clinical measurement of contrast sensitivity and determines the contrast required to read large letters of a fixed size. Total number of letters correctly identified in the affected and fellow eye were reported. The total possible range is 0 to 48. More the number of letters identified, better is the contrast sensitivity.
Time Frame: Weeks 12, 24 and 36
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Placebo: Double-blind Period | Atacicept: Double-blind Period
Number analyzed (Participants) | 15 | 14
letters
  Affected eye: Week 12 (n = 15, 14) | 35.4 (5.9) | 32.4 (8.8)
  Affected eye: Week 24 (n = 5, 5) | 34.2 (6.9) | 33.0 (4.7)
  Affected eye: Week 36 (n = 3, 3) | 37.0 (5.3) | 34.7 (3.2)
  Fellow eye: Week 12 (n = 15, 14) | 38.3 (4.1) | 37.6 (3.3)
  Fellow eye: Week 24 (n = 5, 5) | 36.2 (9.4) | 37.4 (2.4)
  Fellow eye: Week 36 (n = 3, 3) | 39.7 (4.0) | 40.0 (1.0)

9. Secondary Outcome: Contrast Sensitivity: Score Line
Description: Contrast sensitivity was measured using the Pelli-Robson charts with letters arranged in groups of 3. Pelli-Robson chart is used for clinical measurement of contrast sensitivity and determines the contrast required to read large letters of a fixed size. The possible score line range is 0 (visual disability) to 16 (normal contrast sensitivity).
Time Frame: Weeks 12, 24 and 36
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo: Double-blind Period | Atacicept: Double-blind Period
Number analyzed (Participants) | 15 | 14
units on a scale
  Affected eye: Week 12 (n = 15, 14) | 12.1 (1.5) | 10.9 (2.9)
  Affected eye: Week 24 (n = 5, 5) | 11.4 (2.6) | 11.2 (1.6)
  Affected eye: Week 36 (n = 3, 3) | 12.3 (2.1) | 11.7 (1.5)
  Fellow eye: Week 12 (n = 15, 14) | 12.9 (1.5) | 12.7 (1.1)
  Fellow eye: Week 24 (n = 5, 5) | 11.8 (3.3) | 12.4 (0.5)
  Fellow eye: Week 36 (n = 3, 3) | 13.3 (1.2) | 13.3 (0.6)

10. Secondary Outcome: Percentage of Participants Converting to Clinically Definite Multiple Sclerosis (CDMS) Second Clinical Attack
Description: Conversion to CDMS was defined as experiencing a second clinical attack meeting all of the following criteria: (a) Neurological abnormality, either newly appearing or re-appearing, with abnormality specified by both (i) Neurological abnormality separated by at least 30 days from onset of a preceding clinical event, and (ii) Neurological abnormality lasting for at least 24 hours; (b) Absence of fever or known infection (fever with temperature [axillary, orally or intraauricularly] greater than 37.5 degree Celsius/99.5 degree Fahrenheit); (c) Objective neurological impairment, correlating with the participant's reported symptoms, defined as either (i) Increase in at least 1 of the functional systems of the Expanded Disability Status Score (EDSS), or (ii) Increase of the total EDSS score. EDSS assesses disability in 8 functional systems and total score ranges from 0 (normal) to 10 (death due to MS). Percentage of participants converting to CDMS (second clinical attack) was reported.
Time Frame: From baseline (Study Day 1) up to Week 36
Population: ITT population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo: Double-blind Period | Atacicept: Double-blind Period
Number analyzed (Participants) | 17 | 17
percentage of participants | 17.6 | 35.3

ADVERSE EVENTS:
Time Frame: Baseline up to Week 48
Description: ITT population of the double-blind period included all randomized subjects according to their randomized treatment. SFU period population included all randomized participants of double-blind period who participated in the 60-week SFU (N=13,14 for Placebo and Atacicept arms respectively).
Groups:
- Placebo: SFU Period: Participants who received placebo matched to atacicept in double-blind period were included in SFU period (60 weeks) following premature termination of the trial.
- Atacicept: SFU Period: Participants who received atacicept in double-blind period were included in SFU period (60 weeks) following premature termination of the trial.
Arm/Group | Placebo: Double-blind Period | Atacicept: Double-blind Period | Placebo: SFU Period | Atacicept: SFU Period
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17 | 1/13 | 2/14
Other Adverse Events (participants affected / at risk) | 14/17 | 16/17 | 6/13 | 10/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo: Double-blind Period (N=17) | Atacicept: Double-blind Period (N=17) | Placebo: SFU Period (N=13) | Atacicept: SFU Period (N=14)
Bacterial pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 1
Multiple sclerosis (Nervous system disorders) | 0 | 0 | 0 | 1
Myelitis transverse (Nervous system disorders) | 0 | 0 | 0 | 1
Myelitis (Nervous system disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo: Double-blind Period (N=17) | Atacicept: Double-blind Period (N=17) | Placebo: SFU Period (N=13) | Atacicept: SFU Period (N=14)
Injection site reaction (General disorders) | 3 | 11 | 1 | 2
Fatigue (General disorders) | 3 | 3 | 0 | 0
Injection site haematoma (General disorders) | 1 | 3 | 0 | 0
Injection site erythema (General disorders) | 1 | 2 | 0 | 0
Injection site pain (General disorders) | 0 | 2 | 0 | 0
Asthenia (General disorders) | 2 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0
Chest discomfort (General disorders) | 1 | 0 | 0 | 0
Injection site pruritus (General disorders) | 0 | 1 | 0 | 0
Injection site swelling (General disorders) | 1 | 0 | 0 | 0
Pain (General disorders) | 1 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 3 | 2
Chest pain (General disorders) | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 3 | 4 | 0 | 2
Dizziness (Nervous system disorders) | 4 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 1 | 0 | 0
Balance disorder (Nervous system disorders) | 1 | 0 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 1
Muscle contractions involuntary (Nervous system disorders) | 0 | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 1
Optic neuritis (Nervous system disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Tongue disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Aerophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Faecal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting in pregnancy (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 1 | 0 | 2
Influenza (Infections and infestations) | 0 | 2 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 1
Cystitis (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 1
Syphilis (Infections and infestations) | 0 | 0 | 0 | 1
Viral pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 4 | 2 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 1 | 0 | 2
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 1
Tracheal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 2 | 0 | 1
Asthenopia (Eye disorders) | 1 | 0 | 0 | 0
Eye haemorrhage (Eye disorders) | 0 | 1 | 0 | 0
Uhthoff's phenomenon (Eye disorders) | 1 | 0 | 0 | 0
Visual acuity reduced (Eye disorders) | 1 | 0 | 0 | 0
Photopsia (Eye disorders) | 0 | 0 | 1 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 1 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 1 | 0 | 0
Blood glucose increased (Investigations) | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pruritus allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Bundle branch block right (Cardiac disorders) | 1 | 0 | 0 | 0
Ventricular arrhythmia (Cardiac disorders) | 1 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Galactorrhoea (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Bone fissure (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Anaemia of pregnancy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 2
Hypertensive crisis (Vascular disorders) | 0 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Stress urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1
Food allergy (Immune system disorders) | 0 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
The Sponsor voluntarily terminated this trial after observing increased Multiple Sclerosis (MS) disease activity in trial 28063 (ATAMS).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to publishing results, Institution and Principal Investigator (PI) must first provide Sponsor with a copy of proposed publication for review at least 30 days prior to submission. If Institution and PI do not agree to modification, they shall so notify Sponsor and postpone submission for additional 60 days to allow Sponsor to seek legal remedies or file patent applications. There is a need for coordinated approach to any publication of results from sites for any multi-site study.